CLINICAL TRIAL: NCT03863119
Title: An Open-Label, Expanded Access Protocol for Boys With Duchenne Muscular Dystrophy Who Have Completed the Long-Term Extension (VBP15-LTE) or VBP15-004 or VBP15-006 Studies
Brief Title: Expanded Access Protocol for Boys With Duchenne Muscular Dystrophy
Status: Available | Type: Expanded Access
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: VBP15-EAP
Record Dates: First submitted 2019-02-21; First posted 2019-03-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Vamorolone; VBP-15; DMD
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — VBP15 compound

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Vamorolone — 2.0 mg/kg/day, 4.0 mg/kg/day, or 6.0 mg/kg/day at physician discretion

SUMMARY:
The intent of this protocol is to provide continued access to vamorolone for subjects in the United States and Canada who have completed the VBP15-LTE, VBP15- 004, or VBP15-006 protocols (and are thereby ineligible to enroll in another trial of vamorolone therapy), during the time a new drug application for vamorolone is under preparation and review.

DETAILED DESCRIPTION:
Vamorolone will be shipped to the subject's family by the study site. The patient will receive standard of care treatment and procedures for management of DMD. Treating Physicians participating in the expanded access program are required to collect and document any physician, patient, or caregiver reported safety events and report to the Sponsor. The subject's dose of vamorolone may be increased or decreased within a range of 2.0 to 6.0 mg/kg/day (only doses of 2 mg/kg, 4 mg/kg and 6 mg/kg are allowed), given once daily. Administration of vamorolone (taken with an 8 ounce (240 ml) glass of full fat milk, or equivalent high-fat food portion) will be unchanged from the VBP15-LTE, VBP15-004, or VBP15-006 studies. In the absence of safety concerns, and while this Expanded Access protocol is active, vamorolone may be provided indefinitely or until approval, provided that the Treating Physician and family agrees that continued administration of vamorolone is in the best interest of the child.

VBP15-EAP (under IND 118942) has been closed as vamaorolone is approved for marketing in the US VBP15-EAP CANADA has been approved by Health Canada on 11 July 2019 and is currently on-going,but not recruiting

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent or legal guardian has provided written informed consent/HIPAA authorization
* Subject has previously completed at a participating US or Canada study site VBP15-LTE up to and including the Month 24 assessments, OR VBP15-004 up to and including the Week 48 assessments, VBP15-006 up to and including the Week 12 assessment
* Subject and parent/guardian are willing and able to comply with recommended study drug administration plan, and standard of care follow-up and monitoring as recommended by their Treating Physician

Exclusion Criteria:

* Subject had a serious or severe adverse event in study VBP15-LTE or VBP15-004 or VBP15-006 that, in the opinion of the Treating Physician and Sponsor, was probably or definitely related to vamorolone use and precludes safe use of vamorolone for the subject in this expanded access program
* Subject and/or parent/guardian are unable and/or unwilling to comply with regular medical care and follow-up as recommended by their Treating Physician throughout participation in the VBP15-EAP

Sex: Male
Age Groups: Child, Adult, Older Adult
Gender Based: Yes

CONTACTS AND LOCATIONS:
Locations (12):
- United States (6):
  - University of California Davis, Davis, California
  - Nemours Children's Hospital, Orlando, Florida
  - urie Children's Hospital of Chicago, Chicago, Illinois
  - Duke University, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Seattle Children's, Seattle, Washington
- Canada (5):
  - Alberta's Children Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Montreal Childrens Hospital, Montreal, Quebec
- Schneider Chidlren's Medical Center, Petah Tikva, Israel

REFERENCES:
- See also: Vamorolone Phase IIa trial in Duchenne Muscular Dystrophy — http://www.ncbi.nlm.nih.gov/pubmed/30219580